CLINICAL TRIAL: NCT03873259
Title: Burst Wave Lithotripsy (BWL) for the Comminution of Urinary Tract Stones: Intraoperative Evaluation of Safety and Effectiveness
Brief Title: Intraoperative Assessment of of Burst Wave Lithotripsy (BWL)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Indiana University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jonathan Harper, MD, Adjunct Professor, Surgery, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SITE00000349; 5P01DK043881-22 (NIH)
Record Dates: First submitted 2019-03-09; First posted 2019-03-13 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-05

CONDITIONS: Renal Calculi; Ureteral Calculi
MeSH Terms: conditions — Kidney Calculi; Ureteral Calculi

STUDY DESIGN:
Masking Description: Some outcomes assessors will be blinded to the treatment conditions. This will include review of video data for tissue injury.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment Group (Experimental): Subjects in this arm receive the 10-minute burst wave lithotripsy intervention dose during their standard-of-care lithotripsy procedure.
  Interventions: Device: Burst Wave Lithotripsy

INTERVENTIONS:
Device: Burst Wave Lithotripsy — Fragment upper urinary tract stones

SUMMARY:
Burst Wave Lithotripsy (BWL) is a novel method of urinary stone fragmentation that uses multi-cycle bursts of low amplitude ultrasound to induce stone fracture. This is in contrast to traditional extracorporeal shock wave lithotripsy (SWL), which employs a brief single compression/tensile cycle of high amplitude (shock) waves to achieve stone fracture. This is a single-arm feasibility study to test the ability of BWL to comminute (fragment) stones in humans.

DETAILED DESCRIPTION:
This is a two-center, single-arm, feasibility study. The two centers are located within the US and include: University of Washington (UW) School of Medicine and Indiana University (IU) Health Urology Clinic.

The investigative study will be performed in the operating room prior to a standard-of-care (SoC) ureteroscopic (URS) laser lithotripsy procedure. The subject will already be under anesthesia. Stones will be limited to ≤ 12 mm.

The study has one (treatment) arm and is approved to enroll up to 40 subjects (with the intent to treat 20 subjects). All subjects will be treated with the same output parameters for up to a maximum of 10 minutes per stone. The output parameters are nominally defined as:

* 350 kil0Hertz (kHz) acoustic frequency
* 7 MegaPascals (MPa) peak negative pressure
* 20 cycle pulse duration
* 17 Hz pulse repetition frequency

A maximum of 3 stones can be treated per subject.

Safety will be monitored by visual observation of the tissue with an ureteroscopic camera, the self-reported occurrences of adverse events, and occurrences of unplanned emergency department or clinic visits. Fragmentation will be measured by visual observation with an ureteroscopic camera and direct measure of stones removed by basket after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Individuals presenting with at least one kidney stone apparent on CT
* Individuals scheduled for clinical stone removal via ureteroscopy (URS)

Exclusion Criteria:

* Individuals under 18 years of age
* Individuals belonging to a vulnerable group (pregnant, mentally disabled, prisoner, etc.)
* Individuals with uncorrected bleeding disorders or coagulopathies
* Individuals taking a clinically significant anticoagulant dose at the time of the procedure
* Individuals with a calcified abdominal aortic aneurysm or calcified renal artery aneurysm
* Individuals with a solitary kidney
* Individuals with a comorbidity risks which, at the discretion of the physician, would make the patient a poor candidate for the BWL procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Safety - Area of Tissue Injury | Day 0 - the day of the experimental procedure immediately following the acoustic procedure.
  The primary safety endpoint is the area of hemorrhage observed through direct visualization with the ureteroscope.
Effectiveness - Volume of Fragments < 2 mm | Day 0 - the day of the experimental procedure immediately following the acoustic procedure.
  The primary effectiveness endpoint is the volume fraction of stone fragments less than 2 mm relative to the original stone volume.

SECONDARY OUTCOMES:
Safety - Adverse Event Assessment | out to 120 days post-procedure
  The secondary safety outcome is the documented occurrence of all adverse events and comparison of the incidence (rate of occurrence) to the adverse events typically associated with shock wave lithotripsy (SWL) and URS
Effectiveness - Time to Full Comminution | Day 0 - the day of the experimental procedure immediately following the acoustic procedure.
  projected time to full comminution defined as the time at which no fragments would be ≤ 2 mm

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Bailey, PhD, MS, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - IU Health North Hospital, Carmel, Indiana
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] May PC, Kreider W, Maxwell AD, Wang YN, Cunitz BW, Blomgren PM, Johnson CD, Park JSH, Bailey MR, Lee D, Harper JD, Sorensen MD. Detection and Evaluation of Renal Injury in Burst Wave Lithotripsy Using Ultrasound and Magnetic Resonance Imaging. J Endourol. 2017 Aug;31(8):786-792. doi: 10.1089/end.2017.0202. Epub 2017 Jun 16. PMID 28521550
- [Background] Maxwell AD, Cunitz BW, Kreider W, Sapozhnikov OA, Hsi RS, Harper JD, Bailey MR, Sorensen MD. Fragmentation of urinary calculi in vitro by burst wave lithotripsy. J Urol. 2015 Jan;193(1):338-44. doi: 10.1016/j.juro.2014.08.009. Epub 2014 Aug 9. PMID 25111910
- [Derived] Bailey MR, Maxwell AD, Cao S, Ramesh S, Liu Z, Williams JC, Thiel J, Dunmire B, Colonius T, Kuznetsova E, Kreider W, Sorensen MD, Lingeman JE, Sapozhnikov OA. Improving Burst Wave Lithotripsy Effectiveness for Small Stones and Fragments by Increasing Frequency: Theoretical Modeling and Ex Vivo Study. J Endourol. 2022 Jul;36(7):996-1003. doi: 10.1089/end.2021.0714. Epub 2022 Jun 22. PMID 35229652
- [Derived] Harper JD, Metzler I, Hall MK, Chen TT, Maxwell AD, Cunitz BW, Dunmire B, Thiel J, Williams JC, Bailey MR, Sorensen MD. First In-Human Burst Wave Lithotripsy for Kidney Stone Comminution: Initial Two Case Studies. J Endourol. 2021 Apr;35(4):506-511. doi: 10.1089/end.2020.0725. Epub 2020 Nov 5. PMID 32940089
- See also: Sponsor Website — http://www.apl.washington.edu/project/project.php?id=bwl